CLINICAL TRIAL: NCT06887270
Title: Peri-procedural Management of Direct Oral Anticoagulants for Central VENOus Catheters in CAncer Patients With Venous Thromboembolism or Atrial Fibrillation (VENOCAT) Pilot Study
Brief Title: Peri-procedural Management of Direct Oral Anticoagulants for Central VENOus Catheters in CAncer Patients With Venous Thromboembolism or Atrial Fibrillation Pilot Study
Acronym: VENO CAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Helliwell Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-5249
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Anticoagulant-induced Bleeding; Direct Oral Anticoagulant; Cancer; Central Venous Catheter; Periprocedural Complication
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Continued DOAC (Experimental): The continued DOAC group will continue their DOAC peri-procedurally as routine without interruption.
  This management strategy was devised based on the cardiac device insertion studies which found continued AC to be a safe and efficacious strategy for cardiac device insertion, which is procedurally similar to tunneled or port CVC insertion. This is the peri-procedural AC strategy for tunneled or port CVC insertion suggested by the Society of Interventional Radiology guidelines.
  Interventions: Other: Continued DOAC
- Interrupted DOAC (Active Comparator): The interrupted DOAC group will take their last DOAC dose on Day -2, unless their DOAC is Dabigatran and their creatinine clearance is < 50mL/min (Cockcroft-Gault equation), in which their last dose will be on Day -3. The DOAC will be resumed on Day +1. This management strategy was utilized in the PAUSE study and was devised taking into account DOAC half-lives, manufacturer recommendations, and available literature. With this strategy, DOACs would be interrupted for three to four halflives, resulting in minimal residual anticoagulant effect. DOAC interruption is described by number of days rather than hours to allow for a simple pragmatic strategy that would be easy to apply in practice and follow by patients. This strategy was found to be safe and efficacious in the PAUSE and cardiac device insertion studies. This is the peri-procedural AC strategy for tunneled or port CVC insertion suggested by the ISTH.
  Interventions: Other: Interrupted DOAC

INTERVENTIONS:
Other: Continued DOAC — The continued DOAC group will continue their DOAC peri-procedurally as routine without interruption.
  Arms: Continued DOAC
Other: Interrupted DOAC — The interrupted DOAC group will take their last DOAC dose on Day -2, unless their DOAC is Dabigatran and their creatinine clearance is < 50mL/min (Cockcroft-Gault equation), in which their last dose will be on Day -3. The DOAC will be resumed on Day +1.
  Arms: Interrupted DOAC

SUMMARY:
The peri-procedural management of direct oral anticoagulants (DOACs) in persons with cancer (PWC) undergoing tunneled or port central venous catheter (CVC) insertion is a common but understudied clinical problem, with conflicting management advice from guidelines and resultant uncertainty for best practices. Data from prospective studies assessing peri-procedural DOAC management exist; however, these data pertain to procedures in the general population. These management strategies may not be applicable to PWC because (1) although CVC insertion is a low risk, image-guided specialized procedure, (2) PWC are at considerably higher risk of peri-procedural bleeding and thrombosis than non-PWC. It is not surprising, therefore, that guideline recommendations and current practices vary widely. To resolve management uncertainty and establish a standard-of-care, the VENOCAT pilot randomized controlled trial (RCT) is a first step that will assess the feasibility of a definitive trial comparing continued vs. interrupted DOAC management in PWC undergoing tunneled or port CVC insertion. Evidence is needed to standardize clinical practice and reduce the risk of bleeding and thrombotic complications.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with VTE or non-valvular AF on prophylactic or therapeutic dose DOAC
2. Active cancer, defined as diagnosed within the past 6 months; or recurrent, regionally advanced, or metastatic cancer; or for which treatment had been administered within 6 months of port or tunneled CVC insertion; or hematologic cancer not in complete remission
3. Pending elective radiologically guided insertion of tunneled or port CVC
4. Able and willing to adhere to peri-procedural DOAC management plan and follow-up

Exclusion Criteria:

1. Creatinine clearance (Cockcroft-Gault equation) <30 mL/min for Dabigatran, Rivaroxaban, or Edoxaban, and <25mL/min for Apixaban
2. Diagnosis of VTE within 21 days
3. Platelet count < 50 x 10^9/L at time of study entry
4. Concomitant strong inhibitors or inducers to P-glycoprotein and/or CYP-3A4

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  proportion of eligible participants successfully recruited to the study and randomized to a treatment arm

SECONDARY OUTCOMES:
Eligibility rate | 1 year
  proportion of screened patients who are eligible
Intervention adherence | 1 year
  proportion of recruited participants that adhere to the assigned study intervention
DOAC level adherence | 1 year
  proportion of recruited participants that complete DOAC level testing
Retention rate | 1 year
  proportion of recruited participants who attend the follow-up visit
Study completion rate | 1 year
  proportion of recruited participants who completed all study procedures appropriately
Reasons for declining participation | 1 year

OTHER OUTCOMES:
Clinically significant bleeding | 30 days
  composite of major bleeding and clinically relevant non-major bleeding at 30 days
Major bleeding | 30 days
  major bleeding at 30 days
Clinically relevant non-major bleeding | 30 days
  Clinically relevant non-major bleeding at 30 days
Recurrent venous thromboembolism | 30 days
  Recurrent venous thromboembolism in those anticoagulated for VTE at 30 days
Arterial thrombosis | 30 days
  Arterial thrombosis in those anticoagulated for AF at 30 days
All-cause mortality | 30 days
  All-cause mortality at 30 days
DOAC levels | within 2 hours of CVC insertion
  A pre-procedural DOAC level will be drawn by blood sample in all participants on Day 0, within two hours of CVC insertion

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No